CLINICAL TRIAL: NCT02753270
Title: Catheter-directed Foam Sclerotherapy With Tumescence of the Great Saphenous Vein Versus Ultrasound Guided Foam Sclerotherapy: Randomised Controlled Trial
Brief Title: Catheter-directed Foam Sclerotherapy With Tumescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jorgete Barreto dos Santos, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12683
Record Dates: First submitted 2016-04-21; First posted 2016-04-27 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Varicose Vein of Lower Limbs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short catheter (Active Comparator): Twenty-five patients will receive the sclerosant foam by a short catheter 18 G. They will be treated with 3% polidocanol foam prepared with a three-way tap and two plastic disposable syringes, according to Tessari's method.
  Interventions: Procedure: Short catheter
- Long catheter preceded by tumescence (Experimental): Twenty-five patients will be receive foam sclerosant by an angiographic catheter 4 French. They will be treated with 3% polidocanol foam prepared with a three-way tap and two plastic disposable syringes, according to Tessari's method.
  Interventions: Procedure: Long catheter preceded by tumescence

INTERVENTIONS:
Procedure: Short catheter — Ultrasound Guided Foam Sclerotherapy in Great Saphenous Vein, measuring from 6 to 10 mm, with Short Catheter.
  Arms: Short catheter
Procedure: Long catheter preceded by tumescence — Ultrasound Guided Foam Sclerotherapy Transcatheter in Great Saphenous Vein, measuring from 6 to 10 mm, Preceded by Tumescence.
  Arms: Long catheter preceded by tumescence

SUMMARY:
Foam sclerotherapy has been established as another option of treatment for varicose veins of the lower limbs. Its advantages are the application to patients with high surgical risk and immediate return to usual activities. Comparing to laser and radiofrequency, it has lower cost and is less painful. Nevertheless, it requires more re-interventions due to venous recanalization.

DETAILED DESCRIPTION:
The aim of this study is to compare two ultrasound guided foam sclerotherapy (UGFS) techniques to great saphenous vein (GSV) by injecting the sclerosant foam through a short catheter without perivenous tumescence and through a long catheter with saline anesthetic tumescence. Method: selection of 50 patients with primary varicose veins, edema (C3EpAsPr of the CEAP classification) and with GSV measuring 6 - 10 mm, 3 cm below the saphenofemoral junction, identified by ultrasound. The study is taking place at the vascular surgery ambulatory of the University of São Paulo. It is a prospective controlled trial with random allocation in two groups according to the foam sclerosant technique injection. The group 1 will receive the sclerosant foam by a short catheter 18 G and in the group 2 an angiographic catheter 4 Fr. will be used. All patients will be treated with 3% polidocanol foam prepared with a three-way tap and two plastic disposable syringes, according to Tessari's method. The access will be by puncture and its place will depend on the insufficient venous extension. It will be at the level of the knee to treat proximal GSV or at the medial ankle to treat the full length of the vein. In group 2, after inserting the long catheter into the GSV, a saline anesthetic solution will be infiltrated around the insufficient venous segment under ultrasound guidance to reduce its diameter. The long catheter will be continuously flushed with 0.9% saline solution until the foam sclerosant injection. In the cases of treating only the proximal GSV, patients will receive a continuous compression with tourniquet below the knee just before the injection and maintained for 5 minutes thereafter. Then, the tributaries in all 50 patients will be treated by phlebectomy under tumescent local anesthesia. Color-duplex ultrasound follow-up is programmed to 7, 28 and 168 days after the treatment. The first one is to check the possibility of deep venous thrombosis, the second is to verify the occlusion rate and the need of another foam injection. The last ultrasound is to check the final occlusion rate.

Hypothesis: UGFS with long catheter preceded of tumescence has a large occlusion rate of the GSV with monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years;
* patients with varicose veins with edema - CEAP classification C3EpAsPr;
* Great saphenous vein incompetence, segmental and total, with diameter from 6 to 10 mm in proximal thigh, 3 cm from the saphenous femoral junction measured by ultrasound.

Exclusion Criteria:

* Allergy to the sclerosant substance;
* acute deep vein thrombosis or pulmonary thromboembolism;
* local infection in the area of sclerotherapy or severe systemic infection;
* prolonged immobilisation;
* symptomatic patent foramen ovale;
* pregnancy;
* peripheral arterial occlusive disease;
* short saphenous vein incompetence association;
* refusal to sign the consent form;
* nonadherence to outpatient treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Great Saphenous Vein Occlusion Rate | Six months after the intervention
  It will be measured by ultrasound

SECONDARY OUTCOMES:
Quality of Life Change | Six months follow-up after the intervention
  It will be measured by the application of the Aberdeen varicose vein questionnaire
Complications | From the intervention until six months follow-up
  It will be considered:
  * anaphylaxis;
  * superficial thrombophlebitis;
  * deep venous thrombosis;
  * pulmonary embolism;
  * visual disturbances;
  * migraine;
  * transient ischemic attack;
  * tissue necrosis;
  * intra arterial injection;
  * neurological injury;
  * edema;
  * skin pigmentation;
  * skin irritation;
  * burning after the sclerosant injection;
  * retaining clots.

CONTACTS AND LOCATIONS:
Overall Officials: Erasmo S Silva, PhD, Study Chair — São Paulo University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Breu FX, Guggenbichler S, Wollmann JC. 2nd European Consensus Meeting on Foam Sclerotherapy 2006, Tegernsee, Germany. Vasa. 2008 Feb;37 Suppl 71:1-29. PMID 18426039
- [Result] Cavezzi A, Tessari L. Foam sclerotherapy techniques: different gases and methods of preparation, catheter versus direct injection. Phlebology. 2009 Dec;24(6):247-51. doi: 10.1258/phleb.2009.009061. PMID 19952380
- [Result] Gohel MS, Epstein DM, Davies AH. Cost-effectiveness of traditional and endovenous treatments for varicose veins. Br J Surg. 2010 Dec;97(12):1815-23. doi: 10.1002/bjs.7256. Epub 2010 Oct 4. PMID 20922783
- [Result] Parsi K, Exner T, Connor DE, Ma DD, Joseph JE. In vitro effects of detergent sclerosants on coagulation, platelets and microparticles. Eur J Vasc Endovasc Surg. 2007 Dec;34(6):731-40. doi: 10.1016/j.ejvs.2007.07.011. Epub 2007 Oct 4. PMID 17919946
- [Result] Rasmussen LH, Lawaetz M, Bjoern L, Vennits B, Blemings A, Eklof B. Randomized clinical trial comparing endovenous laser ablation, radiofrequency ablation, foam sclerotherapy and surgical stripping for great saphenous varicose veins. Br J Surg. 2011 Aug;98(8):1079-87. doi: 10.1002/bjs.7555. PMID 21725957
- [Result] Coleridge-Smith P, Labropoulos N, Partsch H, Myers K, Nicolaides A, Cavezzi A. Duplex ultrasound investigation of the veins in chronic venous disease of the lower limbs--UIP consensus document. Part I. Basic principles. Eur J Vasc Endovasc Surg. 2006 Jan;31(1):83-92. doi: 10.1016/j.ejvs.2005.07.019. Epub 2005 Oct 14. PMID 16226898
- [Result] Tessari L, Cavezzi A, Frullini A. Preliminary experience with a new sclerosing foam in the treatment of varicose veins. Dermatol Surg. 2001 Jan;27(1):58-60. PMID 11231246
- Available data/document: Study Protocol — http://www.ncbi.nlm.nih.gov/pubmed/18426039
- Available data/document: Study Protocol — http://www.ncbi.nlm.nih.gov/pubmed/19952380
- Available data/document: Literature Review — http://www.ncbi.nlm.nih.gov/pubmed/20922783
- Available data/document: Literature Review — http://www.ncbi.nlm.nih.gov/pubmed/?term=In+vitro+effects+of+detergent+sclerosants+on+coagulation%2C+platelets+and+microparticles.
- Available data/document: Literature Review — http://www.ncbi.nlm.nih.gov/pubmed/21725957
- Available data/document: Literature Review — http://www.ncbi.nlm.nih.gov/pubmed/16226898
- Available data/document: Literature Review — http://www.ncbi.nlm.nih.gov/pubmed/11231246